CLINICAL TRIAL: NCT06143618
Title: The Effect of Education Provided With Escape Room Game and Role Playing Method on Nursing Students' Skills in Evaluating Violence and Their Attitudes Towards Violence
Brief Title: Escape Room Game and Role Playing Method and Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Pinar Akbas, assistant professor doctor, Gazi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: escape room game
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Escape Room Games and Role Playing Gamification
Keywords: escape room games; role playing gamification; violence
MeSH Terms: interventions — Role Playing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- escape room games (Experimental): The escape room game will include a patient scenario of four female patients who are victims of violence and apply to different clinics. Necessary equipment and materials will be provided and stations will be established where four female patients who are victims of violence will be evaluated. In order for them to solve puzzles and puzzles related to the subject at the stations; Colorful puzzle set, lettered chest lock, ballot box, colorful stickers, digital countdown clock, and materials to be used by students will be provided by the researchers. In the game, each student will contact the patient at only one station and evaluate signs and symptoms of violence. The group, which completes the tasks and activities and collects the puzzle pieces that will lead to the code of the lock, will complete the puzzle and enter the number codes on it into the key of the locked box on the table (4 numerical codes received), open the box and get the message 'you can escape'.
  Interventions: Behavioral: escape room games
- role playing (Experimental): In the role play application, there will be scenarios of four female patients who are victims of violence and apply to different clinics. Before the role play activities, students will be asked to form groups of 4-5 people, and each week, a group will be asked to choose one of the four scenarios given by lot and improvise the case-based role play activity within 40 minutes.
  Interventions: Behavioral: role playing
- control (No Intervention): No application will be given to the control group other than theoretical lectures. The theoretical course covers the definition of violence, types of violence, symptoms and findings seen in women exposed to violence, and evaluation of violence. The theoretical course will be delivered in the form of verbal explanation supported by power point presentation. Before the intervention, one week after the intervention and one month later, all students will be administered the Violence Against Women Knowledge Test, the Attitudes towards Violence Scale and the Scale for Nurses and Midwives to Recognize the Signs of Violence Against Women.

INTERVENTIONS:
Behavioral: escape room games — The escape room game will include a patient scenario of four female patients who are victims of violence and apply to different clinics. Necessary equipment and materials will be provided and stations will be established where four female patients who are victims of violence will be evaluated. In the game, each student will contact the patient at only one station and evaluate signs and symptoms of violence. The activities at the stations will be carried out together as a group. The group, which completes the tasks and activities and collects the puzzle pieces that will lead to the code of the lock, will complete the puzzle and enter the number codes on it into the key of the locked box on the table (4 numerical codes received), open the box and get the message 'you can escape'. The group with the most time left at the end of the game will come first and will be rewarded.
  Arms: escape room games
Behavioral: role playing — In the role play application, there will be scenarios of four female patients who are victims of violence and apply to different clinics. Before the role play activities, students will be asked to form groups of 4-5 people, and each week, a group will be asked to choose one of the four scenarios given by lot and improvise the case-based role play activity within 40 minutes. Before the role play application, the materials that may be required for the students (clothes, materials, etc.) and the preparation of the environment (hospital, polyclinic, etc.) will be provided by the researchers in accordance with the activity to be enacted. At the end of the role play activities, students will be able to express, evaluate and discuss their feelings and thoughts within and between groups.
  Arms: role playing

SUMMARY:
In this regard, we think that escape room games and role playing gamification methods used in nursing education can be effective in gaining these skills. For this reason, we aim to evaluate the effect of training on diagnosing and evaluating violence against women, given using escape room game and role-playing methods, on nursing students' skills in diagnosing and evaluating violence against women and their attitudes towards violence. The research is a pre-test-post-test randomized controlled, factorial group experimental study.

DETAILED DESCRIPTION:
Violence is a social problem where a person uses physical, social, psychological, sexual, emotional and economic power over another person and has negative effects on the person. According to the person exposed, violence against women, children, elderly people, disabled people, LGBT individuals, and immigrants is grouped as violence among peers. Violence refers to the physical damage that can be directly perceived by outside observers or medically detectable by health professionals, as well as the psychological damage that these individuals experience, which are difficult to notice or show unnoticed psychosomatic symptoms. In this context, nurses face many difficulties in the process of diagnosing, evaluating and preventing violence in the provision of health services, which prevent intervention, such as not being able to recognize cases of violence, remaining indifferent, not considering such cases within the scope of their professional responsibilities, or not having sufficient knowledge and skills, and feeling inadequate in the care of forensic cases. In nursing education, in addition to imparting theoretical knowledge about violence to students, it is necessary to provide basic clinical skills such as effective communication skills with individuals exposed to violence, cognitive skills and technological skills.

Gamification is a method used to improve problem-solving skills by reasoning in the presentation of information and to ensure that learning becomes permanent by arousing excitement and curiosity. Particularly, the use of gamification in the education process makes the teaching-learning process more attractive, increases students' motivation, and allows students to develop interesting skills. Various methods are suggested to increase students' participation in the gamification process. Examples of innovative approaches used in the gamification process are escape room games and role-playing games. Role-play, which is an active teaching method, is a method that enables nurses to play a role in an environment similar to the clinical environment, which can help them prepare to face real cases in the clinical environment and enables learning by playing. Role playing is used as a skill-focused teaching method that provides social communication skills, active listening, empathy of emotions, and seeing sections from real life in teaching knowledge and skills in education, and is among the educational methods used to raise awareness in nursing. In the escape room game, in problem-based learning, a problem is presented and students must investigate it and offer possible solutions. The premise of an escape room is that a group of participants work collaboratively using clues that include puzzles and specific objectives to "escape" the room before they run out of time to solve a problem.

The basis of nursing education, in addition to transferring theoretical knowledge, is to provide nursing students with skills such as critical thinking, problem-solving skills, decision-making, holistic care, effective communication and teamwork. In the context of nursing education and training, escape rooms and role-playing games allow students to use the latest technological developments, solve both physical and mental puzzles or tests, acquire basic professional competencies, develop teamwork skills, and use multiple intelligences to solve problems. In this context, researchers think that escape room games and role-playing gamification methods used in nursing education may be effective in gaining these skills. Therefore, it is aimed to evaluate the effect of training on diagnosing and evaluating violence against women, given using escape room games and role-playing methods, on nursing students' skills in diagnosing and evaluating violence against women and their attitudes towards violence.

ELIGIBILITY:
Inclusion Criteria:

* Registering for the Obstetrics and Gynecology Nursing course for the first time,
* Volunteering to participate in the research.

Exclusion Criteria:

* Having a high school, associate or bachelor's degree in a health-related field,
* Having difficulty in understanding and speaking Turkish.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Information on violence against women | Change in initial violence information in one week and one month
  Measurements will be made using the Violence Against Women Knowledge Test. The lowest score that can be obtained from the test is 0 and the highest score is 100. As the score obtained from the test increases, the level of knowledge increases.
Attitude towards violence | Change in initial attitude towards violence in 1 week and 1 month
  Measurements will be made using the Attitudes Towards Violence Scale. The average attitude score that can be obtained from the scale varies between 19 and 95. A high attitude score indicates an increase in traditionalism in the attitude of healthcare personnel towards violence, while a low attitude score indicates a move away from tradition and a contemporary view.
Recognizing signs of violence | change in recognition of signs of violence at baseline, at 1 week, and at 1 month
  Measurements will be made using the Scale for Nurses and Midwives to Recognize Signs of Violence Against Women. The highest score to be obtained from the scale is "31" and the lowest score is "0". A high score indicates that the level of knowledge regarding recognizing the signs of violence against women is sufficient.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan ÖZKAN ŞAT, PhD, Principal Investigator — Bitlis Eren University; Nurhan AKTAŞ, PhD, Principal Investigator — Sakarya University
Locations (2):
- Turkey (Türkiye) (2):
  - Bitlis Eren University Faculty of Health Sciences, Bitlis
  - Karabük University Faculty of Health Sciences, Karabük

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR